CLINICAL TRIAL: NCT02498418
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multicenter, Bioequivalence Study With Clinical Endpoint Comparing Rifaximin 200-mg Tablets With Xifaxan® 200-mg Tablets in the Treatment of Travelers' Diarrhea
Brief Title: Study Comparing Rifaximin With Xifaxan 200 mg in Traveler's Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACTA/RIFX/2015
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Generic Rifaximin 200 mg Tablets (Experimental): Participants will receive a generic rifaximin 200 mg tablet 3 times daily orally for 3 days.
  Interventions: Drug: Rifaximin
- Xifaxan 200 mg Tablets (Active Comparator): Participants will receive a xifaxan 200 mg tablet 3 times daily orally for 3 days.
  Interventions: Drug: Xifaxan®
- Placebo (Placebo Comparator): Participants will receive a rifaximin placebo tablet 3 times daily orally for 3 days.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Rifaximin — Tablets, generic formulation of the brand product.
  Arms: Generic Rifaximin 200 mg Tablets
Drug: Xifaxan® — Tablets, brand product.
  Arms: Xifaxan 200 mg Tablets
Drug: Placebo Tablet — Placebo tablets in the same image of the generic rifaximin. Has no active ingredient.
  Arms: Placebo

SUMMARY:
The primary objective is to demonstrate rifaximin 200 milligrams (mg) tablets (test) and Xifaxan® 200 mg tablets (reference) are clinically bioequivalent with respect to the clinical cure rates when administered 3 times a day (TID) for 3 days in participants with travelers' diarrhea.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled bioequivalent study with a clinical endpoint in the treatment of travelers' diarrhea. After 3 unformed stools are recorded within the 24 hours immediately preceding randomization, participants are to be randomized to receive the generic rifaximin 200 mg oral tablet, Xifaxan (the reference listed drug)200 mg oral tablet, or placebo 3 times daily for 3 days (that is; on Days 1, 2, and 3).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or nonpregnant female aged ≥18 years non-indigenous travelers (for example; visiting students/faculty or international tourists) affected by naturally acquired acute diarrhea. Diarrhea is defined as the passage of at least 3 unformed stools in a 24-hour period. Stools are classified as formed (retains shape), soft (assumes shape of container), or watery (can be poured). When using this classification, both soft and watery stools are unformed and abnormal.
2. At least 3 unformed stools recorded within the 24 hours immediately preceding randomization.
3. At least 1 of the following signs and symptoms of enteric infection:

   * abdominal pain or cramps
   * nausea
   * vomiting
   * fecal urgency
   * excessive gas/flatulence
   * tenesmus
4. Women of child-bearing potential have a negative pregnancy test prior to beginning therapy and agree to use effective contraceptive methods during the study.

Exclusion Criteria:

1. Pregnant, breast feeding, or planning a pregnancy.
2. Immediately prior to randomization, acute diarrhea for >72 hours.
3. Presence of:

   * fever (≥100 degrees fahrenheit [°F] or ≥37.8 degrees celsius [°C]), or
   * hematochezia (blood in stool), or
   * clinical findings suggesting moderate or severe dehydration.
4. Active, uncontrolled, or clinically significant diseases or disorders of the heart, lung, kidney, gastrointestinal (GI) tract (other than infectious diarrhea in travelers), or central nervous system.
5. Administration of any of the following:

   * any antimicrobial agents with an expected activity against enteric bacterial pathogens within 7 days preceding randomization
   * more than 2 doses of a symptomatic antidiarrheal compound such as antimotility agents, absorbent agents, and antisecretory agents within 8 hours preceding randomization
6. Use of any drug such as aspirin or ibuprofen (Advil), which can cause GI bleeding. Acetaminophen (Tylenol) or paracetamol is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Actavis Inc.
Locations (1):
- Site 1, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 739 nonindigenous travelers with naturally acquired acute diarrhea were enrolled and randomized in this study.
Groups:
- Generic Rifaximin 200 mg Tablets: Participants received a generic rifaximin 200 milligrams (mg) tablet 3 times daily orally for 3 days.
- Xifaxan 200 mg Tablets: Participants received a xifaxan 200 mg tablet 3 times daily orally for 3 days.
- Rifaximin Placebo Tablets: Participants received a rifaximin placebo tablet 3 times daily orally for 3 days.
Period: Overall Study
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets
Started | 247 | 248 | 244
Safety Population (Received at least 1 dose of study drug.) | 246 | 247 | 244
Modified Intent-to-treat Population (Met inclusion/exclusion criteria, took ≥1 dose of study drug, provided efficacy and safety data.) | 183 | 186 | 180
Per-protocol Analysis Set (Met study criteria, completed Visit 3 within 24-72 hrs of last dose, had no major protocol violation) | 182 | 181 | 176
Completed | 245 | 246 | 238
Not Completed | 2 | 2 | 6
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Participant taken prohibited medication | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population included all the participants who satisfied the inclusion and exclusion criteria and were randomized into the study.
Groups:
- Generic Rifaximin 200 mg Tablets: Participants received a generic rifaximin 200 mg tablet 3 times daily orally for 3 days.
- Total: Total of all reporting groups
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets | Total
Number analyzed (Participants) | 247 | 248 | 244 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (15.78) | 44.3 (16.58) | 42.0 (15.21) | 42.9 (15.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 130 | 132 | 385
  Male | 124 | 118 | 112 | 354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 189 | 188 | 188 | 565
  Not Hispanic or Latino | 58 | 58 | 54 | 170
  Unknown or Not Reported | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 18 | 13 | 54
  White | 208 | 222 | 220 | 650
  More than one race | 13 | 5 | 9 | 27
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Cure at Test of Cure (TOC) Visit (Within 24 to 72 Hours From the Time of Last Dose): Per-Protocol (PP) Population
Description: Clinical cure was defined as either of the following: No stools or only formed stools within a 48-hour period and no fever, with or without other enteric symptoms or; No watery stools or no more than 2 soft stools passed within a 24-hour period with no fever and no other enteric symptoms except for mild excess gas/flatulence. Bioequivalence evaluation between test (generic rifaximin 200 mg tablets) and reference groups (xifaxan 200 mg tablets) was conducted in this endpoint, hence placebo group was not included. Participants who were discontinued early from the study due to lack of treatment effect after completing 9 doses within 72 hours from the time of first dose were included in the PP population using Last Observation Carried Forward (LOCF) method. Additionally, participants whose condition worsened and who required alternate or supplemental therapy for the treatment of travelers' diarrhea were discontinued and included in the PP population analysis using LOCF.
Time Frame: TOC visit (Day 5, 6 or 7)
Population: PP population: randomized participants, met inclusion/exclusion criteria, took 3 days of study drug, were compliant with study drug dose, and completed Visit 3 within 24-72 hours from the time of last dose, with no major protocol deviations/violations that would affect treatment evaluation. LOCF method was used as applicable for this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets
Number analyzed (Participants) | 182 | 181
Participants | 90 | 93
Statistical Analysis 1: Comparison: Generic Rifaximin 200 mg Tablets vs Xifaxan 200 mg Tablets; Bioequivalence was evaluated based on the PP analysis set using Z-test with Yates correction; Test type: Equivalence — Bioequivalence was demonstrated if 90% confidence interval (CI) of percentage difference between generic rifaximin 200 mg tablets and xifaxan 200 mg tablets was within the equivalence range (-20%, +20%); Difference in percentage of participants = -0.0193, 90% CI 2-sided [-0.11 to 0.07]

2. Secondary Outcome: Time to Last Unformed Stool (TLUS)
Description: TLUS was defined as the interval beginning with the first dose of study drug and ending with the last unformed stool passed within a period of 120 hours (within 48 hours from the time of last dose [at 72 hours]). Mathematically, TLUS was calculated as follows. TLUS (hours) = date/time of last unformed stool within 48 hours from the time of last dose - date/time of first dose.
Time Frame: Day 1 to Day 5
Population: mITT population included all randomized participants who met all inclusion and none of the exclusion criteria, received at least 1 dose of study drug and provided efficacy and safety data after 1 dose of study drug. Here, 'Overall number of participants analyzed'=participants with TLUS in the mITT population.
Measure: Median (Full Range); unit: hours
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets
Number analyzed (Participants) | 182 | 186 | 178
hours | 65.25 [3.93 to 119.42] | 65.75 [14.10 to 117.08] | 67.01 [16.65 to 117.87]

3. Secondary Outcome: Percentage of Participants Who Achieved Microbiological Cure at TOC Visit (Within 24 to 72 Hours From the Time of Last Dose)
Description: Participants were considered to have achieved microbiological cure if the pathogen identified at Day 1 is no longer found in the stool at the TOC visit.
Time Frame: TOC visit (Day 5, 6, or 7)
Population: mITT population: all randomized participants who met all inclusion and none of the exclusion criteria, received at least 1 dose of study drug and provided efficacy and safety data after 1 dose. 'Overall number of participants analyzed'=participants evaluable for this endpoint. 'Number analyzed'=participants evaluable for the specified categories.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets
Number analyzed (Participants) | 51 | 47 | 46
percentage of participants
  Escherichia coli | 25.5 | 31.9 | 17.4
  Enterotoxigenic Escherichia coli (ETEC): number analyzed (Participants) | 23 | 22 | 19
  Enterotoxigenic Escherichia coli (ETEC) | 43.5 | 54.5 | 68.4
  Enteroaggregative Escherichia coli (EAEC): number analyzed (Participants) | 25 | 22 | 23
  Enteroaggregative Escherichia coli (EAEC) | 32.0 | 27.3 | 26.1
  Other microorganisms: number analyzed (Participants) | 17 | 22 | 14
  Other microorganisms | 70.6 | 81.8 | 92.9
  Stool microscopy for ova and parasites: number analyzed (Participants) | 6 | 3 | 5
  Stool microscopy for ova and parasites | 83.3 | 100.0 | 100.0

4. Primary Outcome: Number of Participants Who Achieved Clinical Cure at TOC Visit (Within 24 to 72 Hours From the Time of Last Dose): Modified Intent-to-Treat (mITT) Population
Description: Clinical cure was defined as either of the following: No stools or only formed stools within a 48-hour period and no fever, with or without other enteric symptoms or; No watery stools or no more than 2 soft stools passed within a 24-hour period with no fever and no other enteric symptoms except for mild excess gas/flatulence. Participants discontinued early for reasons other than "lack of treatment effect after completing 9 doses within 72 hours from the time of first dose" and for "participants whose condition worsened and who required alternate or supplemental therapy for the treatment of travelers' diarrhea" were included in the mITT population analysis using LOCF.
Time Frame: TOC visit (Day 5, 6 ,or 7)
Population: mITT population included all randomized participants who met all inclusion and none of the exclusion criteria, received at least 1 dose of study drug and provided efficacy and safety data after 1 dose of study drug. LOCF method was used as applicable for this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets
Number analyzed (Participants) | 183 | 186 | 180
Participants | 91 | 95 | 86
Statistical Analysis 1: Comparison: Generic Rifaximin 200 mg Tablets vs Rifaximin Placebo Tablets; 95% CIs was calculated using Z-test with Yates' correction; Test type: Superiority; p = 0.7899, Z-test — Threshold of significance at 0.05 level; Difference in percentage of participants = -0.0195, 95% CI 2-sided [-0.09 to 0.13]
Statistical Analysis 2: Comparison: Xifaxan 200 mg Tablets vs Rifaximin Placebo Tablets; 95% CIs was calculated using Z-test with Yates' correction; Test type: Superiority; p = 0.5987, Z-test — Threshold for significance at 0.05 level; Difference in percentage of participants = 0.0330, 95% CI 2-sided [-0.07 to 0.14]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 7
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Generic Rifaximin 200 mg Tablets | Xifaxan 200 mg Tablets | Rifaximin Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/246 | 0/247 | 0/244
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/247 | 0/244
Other Adverse Events (participants affected / at risk) | 17/246 | 17/247 | 24/244
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Rifaximin 200 mg Tablets (N=246) | Xifaxan 200 mg Tablets (N=247) | Rifaximin Placebo Tablets (N=244)
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Defecation urgency (Gastrointestinal disorders) | 1 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 4 | 3 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Rectal tenesmus (Gastrointestinal disorders) | 3 | 4 | 8
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Urine leukocyte esterase (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02498418/SAP_000.pdf
  • Study Protocol (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT02498418/Prot_001.pdf